CLINICAL TRIAL: NCT07018882
Title: Single-Center, Single-arm, Open, Prospective, Pivotal Clinical Trial for Evaluating the Audiological Efficacy and Safety of Sullivan Cochlear Implantation in Patients With Severe to Profound Bilateral Hearing Loss.
Brief Title: Evaluation of the Efficacy and Safety of the Sullivan Cochlear Implant.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Todoc (Industry)
Collaborators: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sullivan
Record Dates: First submitted 2025-05-22; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Hearing Loss, Sensorineural
Keywords: cochlear implant
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sullivan (Experimental)
  Interventions: Device: Sullivan

INTERVENTIONS:
Device: Sullivan — Patients who are clinically eligible for cochlear implant surgery and can tolerate the surgery will be asked for their consent and then undergo the cochlear implant procedure. The outcome of the cochlear implant surgery will be evaluated through auditory performance assessments. Additionally, adverse effects will be monitored to assess the efficacy and safety of the cochlear implants on auditory function.

SUMMARY:
The study will be conducted as a prospective, single center, repeat measure, single-arm, open label clinical study

DETAILED DESCRIPTION:
This study is a clinical trial designed to examine the auditory performance improvement in patients with bilateral severe sensorineural hearing loss (70 dB HL or greater) by comparing auditory performance before and after cochlear implant surgery.

Cochlear implants, both imported and domestically manufactured, have already been approved and are in use in the country. These existing devices have also undergone clinical research, comparing and analyzing auditory performance before and after implantation. Therefore, this study is designed as a prospective, single-arm, open-label clinical trial.

Patients who are clinically eligible for cochlear implant surgery and can tolerate the surgery will be asked for their consent and then undergo the cochlear implant procedure. The outcome of the cochlear implant surgery will be evaluated through auditory performance assessments.

Additionally, adverse effects will be monitored to assess the efficacy and safety of the cochlear implants on auditory function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sensorineural hearing loss of 1 side or both sides (70 dBHL) or higher, aged 19 years or older
* No previous cochlear implantation history in the ear scheduled for surgery
* No contraindications to surgery, such as cochlear agenesis or auditory nerve agenesis, as determined by imaging tests
* Patients without cancer, autoimmune disease, or neurological disease
* Patients with a general condition that allows general anesthesia
* Patients with no abnormalities in personality, depression, anxiety, sociality, or problem drinking tests
* Use Korean
* Patients who agree to participate in the clinical trial and sign a written consent form However, if the patient is unable to sign, the patient (if able to sign) and guardian (or agent) voluntarily agree to participate in the clinical trial and sign an informed consent form

Exclusion Criteria:

* Cases where electrode insertion is difficult due to severe internal malformation, cochlear ossification, etc.
* Cases with cancer or autoimmune disease
* Cases with a general condition that makes it difficult to tolerate general anesthesia
* Cases with moderate or higher mental disability or where auditory training is difficult due to the absence of parents or supporters to assist with rehabilitation education
* Cases deemed inappropriate for this test by the clinical trial manager

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in open-set sentence recognition | at 12-week and 24-week post-implant
  Sentences will be presented before the implant surgery, and at 12- and 24-weeks post implant, to assess and record the patient's sentence recognition ability. A total of 10 sentences, comprising 50 words, will be used for this evaluation.
  For each sentence, the percentage of correctly recognized words will be calculated out of the total 50 words across the 10 sentences. Sentence recognition abilities for each participant will be assessed at pre-surgery, 12 weeks, and 24 weeks. Improvement in sentence recognition at 12 weeks and 24 weeks will be determined by comparing these post-implant scores with pre-surgery scores.

SECONDARY OUTCOMES:
Change in open-set monosyllabic word recognition | at the 12-week and 24-week post-implant
  Pre- and post-implant (at 12 and 24 weeks) monosyllabic word recognition will be assessed by presenting words auditorily, with results recorded, compared, and observed. The assessment will use 20 monosyllabic words.
  For each participant, pre-surgery, 12-week, and 24-week monosyllabic word recognition scores will be calculated as the percentage of correctly recognized words out of the total 20 words.
  The difference in monosyllabic word recognition between pre-surgery and 12 weeks post-surgery, as well as between pre-surgery and 24 weeks post-surgery, will be calculated.
Change in open-set bisyllabic word recognition | at the 12-week and 24-week post-implant
  Pre- and post-implant (at 12 and 24 weeks) bisyllabic word recognition will be assessed by presenting words auditorily, with results recorded, compared, and observed. The cognitive assessment will use 20 bisyllabic words.
  For each participant, pre-surgery, 12-week, and 24-week bisyllabic word recognition scores will be calculated as the percentage of correctly recognized words out of the total 20 words.
  The difference in bisyllabic word recognition between pre-surgery and 12 weeks post-surgery, as well as between pre-surgery and 24 weeks post-surgery, will be calculated.
Change in pure-tone hearing thresholds | at the 12-week and 24-week post implant
  The average minimum pure-tone hearing thresholds before and after implant surgery (at 12 and 24 weeks) will be compared and observed.
  The average minimum pure-tone hearing threshold is calculated as the mean of the minimum hearing thresholds at 500, 1000, 2000, and 3000 Hz.